CLINICAL TRIAL: NCT04898270
Title: Clinical Efficacy and Benefit of Reducing Metabolic Syndrome by Adjunctive Use of Fute (Flupentixol) in Multi-acting Receptor-targeted Antipsychotics (MARTAs) Treated Schizophrenia Patients
Brief Title: Adjunctive Use of Fute (Flupentixol) in Multi-acting Receptor-targeted Antipsychotics Treated Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SG19331B
Record Dates: First submitted 2021-04-23; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia; Psychosis; Metabolic Syndrome; Flupentixol; Antipsychotic Agents; Central Nervous System Diseases; Clinical Therapy; Olanzapine; Quetiapine
Keywords: Schizophrenia; Metabolic Syndrome; Flupentixol; olanzapine; quetiapine; Central Nervous System Diseases; Clinical Therapy; Antipsychotic Agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Metabolic Syndrome; Central Nervous System Diseases | interventions — Flupenthixol

STUDY DESIGN:
Intervention Model Description: It is expected to be admitted to patients with schizophrenia who are over 20 years old and are being treated with MARTAs antipsychotics due to poor treatment efficacy or significant weight gain after use, poor blood sugar control, and other metabolic syndrome-related problems, but Patients who do not meet the medication standards for diabetes or hyperlipidemia, and are willing to accept additional use of Flupentixol after evaluation by the physician.
  To compare whether the original MARTAs dose can be effectively reduced after additional use of Flupentixol for at least 12 weeks, whether the symptoms of psychosis have improved, and whether the various factors of metabolic syndrome have improved.
Who Masked: Participant
Masking Description: It is expected to be admitted to patients with schizophrenia who are over 20 years old and are being treated with MARTAs antipsychotics due to poor treatment efficacy or significant weight gain after use, poor blood sugar control, and other metabolic syndrome-related problems, but Patients who do not meet the medication standards for diabetes or hyperlipidemia, and are willing to accept additional use of Flupentixol after evaluation by the physician.
  To compare whether the original MARTAs dose can be effectively reduced after additional use of Flupentixol for at least 12 weeks, whether the symptoms of psychosis have improved, and whether the various factors of metabolic syndrome have improved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MARTAs combined with flupentixol (Experimental): Flupentixol tablets are indicated for:
  • maintenance therapy of chronic schizophrenic patients whose main manifestations do not include excitement, agitation, or hyperactivity.
  Other Names:
  Fute tables, Fluanxol
  Multi-acting receptor-targeted antipsychotics (MARTAs): clozapine, olanzapine, quetiapine.
  Interventions: Drug: Flupentixol; Drug: Multi-acting receptor-targeted antipsychotics (MARTAs)
- Multi-acting receptor-targeted antipsychotics (MARTAs) (Active Comparator): clozapine, olanzapine, quetiapine
  Interventions: Drug: Multi-acting receptor-targeted antipsychotics (MARTAs)

INTERVENTIONS:
Drug: Flupentixol — Flupentixol tablets are indicated for:
  • maintenance therapy of chronic schizophrenic patients whose main manifestations do not include excitement, agitation, or hyperactivity.
  Other Names: Fute tables; Fluanxol
  Arms: MARTAs combined with flupentixol
Drug: Multi-acting receptor-targeted antipsychotics (MARTAs) — Multi-acting receptor-targeted antipsychotics (MARTAs)

SUMMARY:
Fute (Flupentixol) combined with MARTAs (Multiple-Acting Receptor Targeted Antipsychotics) drugs has its clinical efficacy toward positive symptoms and might reduce the metabolic syndrome-related factors in patients. This study is the first clinical trial to explore the treatment of patients with flupentixol combined with MARTAs. However, due to research limitations, the number of patients who participated in the clinical trial is small, and it depends on subsequent larger-scale clinical trials for more in-depth verification.

DETAILED DESCRIPTION:
Objectives

The effects of adjunctive Fute (Flupentixol) with MARTAs (Multiple-Acting Receptor Targeted Antipsychotics) on the metabolic profiles of patients and clinical efficacy of treatment in schizophrenia.

Methodology

It is expected to be admitted to patients with schizophrenia who are over 20 years old and are being treated with MARTAs antipsychotics due to poor treatment efficacy or significant weight gain after use, poor blood sugar control, and other metabolic syndrome-related problems, but Patients who do not meet the medication standards for diabetes or hyperlipidemia, and are willing to accept additional use of Flupentixol after evaluation by the physician.

To compare whether the original MARTAs dose can be effectively reduced after additional use of Flupentixol for at least 12 weeks, whether the symptoms of psychosis have improved, and whether the various factors of metabolic syndrome have improved.

Number of patients

It is estimated that 30 subjects will be recruited to participate in this clinical trial. This report is an interim report with the results of 15 subjects.

Diagnosis and main criteria for inclusion

Patients suffering from schizophrenia who are over 20 years old and are using MARTAs antipsychotics.

Test product, dose and mode of administration, batch number

Fute F.C. Tablets (Flupentixol), the clinically recommended dosage should be adjusted according to the individual conditions of the patients. Generally speaking, a low dose should be administered at the beginning. Then the dosage is increased according to the treatment response to achieve the appropriate curative effect as soon as possible. The maintenance dose is usually administered as a single dose in the morning, and the maintenance dose is usually 5-20 mg/day.

The initial dose is 3-15 mg/day, divided into 2-3 administrations, and can be increased to 40 mg/day if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from schizophrenia are over 20 years old and are using MARTAs antipsychotics.

Exclusion Criteria:

* >65y aged Patients.
* >Other non-schizophrenia disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Severity scale (CGI-S) | 12 weeks
  The clinical efficacy of schizophrenia, Clinical Global Impression-Severity scale (CGI-S), in patients taking MARTAs combined with Flupentixol for 12 weeks.
  The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.
  CGI-Severity (CGI-S) which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  This rating is based upon observed and reported symptoms, behavior, and function in the past seven days.
Positive and Negative Syndrome Scale (PANSS) | 12 weeks
  The clinical efficacy of schizophrenia, Positive and Negative Syndrome Scale (PANSS), in patients taking MARTAs combined with Flupentixol for 12 weeks.
  PANSS is a medical scale used for measuring symptom severity of patients with schizophrenia. It is widely used in the study of antipsychotic therapy. The scale is known as the "gold standard" that all assessments of psychotic behavioral disorders should follow.
  The name refers to the two types of symptoms in schizophrenia, as defined by the American Psychiatric Association: positive symptoms, which refer to an excess or distortion of normal functions (e.g., hallucinations and delusions), and negative symptoms, which represent a diminution or loss of normal functions. Some of these functions which may be lost include normal thoughts, actions, ability to tell fantasies from reality, and the ability to properly express.

SECONDARY OUTCOMES:
Fasting blood glucose (FBG) in mg/dL | 12 weeks
  Metabolic syndrome-related factors in patients, fasting blood glucose in mg/dL
Cholesterol in mg/dL | 12 weeks
  Metabolic syndrome-related factors in patients, cholesterol in mg/dL
High-density lipoprotein (HDL) cholesterol in mg/dL | 12 weeks
  Metabolic syndrome-related factors in patients, high-density lipoprotein (HDL) cholesterol in mg/dL
Low-density lipoprotein (LDL) cholesterol in mg/dL | 12 weeks
  Metabolic syndrome-related factors in patients, low-density lipoprotein (LDL) cholesterol in mg/dL
Blood creatinine in mg/dL | 12 weeks
  Metabolic syndrome-related factors in patients, blood creatinine in mg/dL
Triglyceride in mg/dL | 12 weeks
  Metabolic syndrome-related factors in patients, triglyceride in mg/dL
Glutamine transaminase (r-GT) in U/L | 12 weeks
  Metabolic syndrome-related factors in patients, glutamine transaminase (r-GT) in U/L
Aspartate transaminase (GOT) in U/L | 12 weeks
  Metabolic syndrome-related factors in patients, aspartate transaminase (GOT) in U/L
Alanine transaminase (GPT) in U/L | 12 weeks
  Metabolic syndrome-related factors in patients, alanine transaminase (GPT) in U/L

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jui Tsai, M.D., Principal Investigator — Taichung Veterans General Hospital (TVGH), Taiwan
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Consider patient privacy.